CLINICAL TRIAL: NCT03202836
Title: Vaginal Progesterone Supplementation in the Management of Preterm Labor: A Randomized, Double Blind, Controlled Trial
Brief Title: Vaginal Progesterone Supplementation in the Management of Preterm Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Vorapong Phupong, Head of Placental Related Diseases Research Unit, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 230/2017
Record Dates: First submitted 2017-06-24; First posted 2017-06-29 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Preterm Labor
MeSH Terms: conditions — Obstetric Labor, Premature | interventions — Progesterone; Utrogestan; Tocolytic Agents; Steroids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vaginal progesterone (Experimental): Vaginal utrogestan 400 mg, vaginal suppository, once at bed time until gestational age 37 weeks and tocolysis plus corticosteroid for 48 hours
  Interventions: Drug: progesterone; Drug: Tocolytics; Drug: Steroids
- no medication (Other): only tocolysis plus corticosteroid for 48 hours
  Interventions: Drug: Tocolytics; Drug: Steroids

INTERVENTIONS:
Drug: progesterone — vaginal utrogestan
  Other Names: utrogestan
  Arms: vaginal progesterone
Drug: Tocolytics — tocolysis for 48 hours
Drug: Steroids — antenatal corticosteroids for 48 hours

SUMMARY:
This study evaluates the addition of vaginal progesterone in the management of preterm labor. Half of participants will receive vaginal progesterone, tocolysis and corticosteroid, while the other half will receive only tocolysis and corticosteroid.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnant women with preterm labor, gestational age 24-34 weeks

Exclusion Criteria:

* have indicated preterm birth
* allergy to progesterone
* fetal anomalies
* cervical dilate > 5 cm.
* have medical disease
* have obstetric complication

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2017-06-29 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Time from preterm labor pain to delivery | 9 weeks
  time since preterm labor to delivery

SECONDARY OUTCOMES:
gestational age at delivery | 9 weeks
  gestational age at birth
number of pregnant women deliver before 34 weeks | 6 weeks
  preterm birth < 34 weeks
number of pregnant women deliver before 37 weeks | 9 weeks
  preterm birth < 37 weeks
Number of newborn with respiratory distress syndrome | 9 weeks
  Number of newborn with respiratory distress syndrome
Number of newborn with intraventricular hemorrhage | 9 weeks
  Number of newborn with intraventricular hemorrhage
Number of newborn with necrotizing enterocolitis | 9 weeks
  Number of newborn with necrotizing enterocolitis
Number of newborn with sepsis | 9 weeks
  Number of newborn with sepsis

CONTACTS AND LOCATIONS:
Overall Officials: Vorapong Phupong, MD, Study Director — Chulalongkorn University
Locations (1):
- Faculty of Medicine, Chulalongkorn University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] O'Brien JM. Vaginal progesterone prophylaxis for preterm birth. Lancet. 2016 Sep 17;388(10050):1159-60. doi: 10.1016/S0140-6736(16)31614-2. Epub 2016 Sep 16. No abstract available. PMID 27650091
- [Background] Azargoon A, Ghorbani R, Aslebahar F. Vaginal progesterone on the prevention of preterm birth and neonatal complications in high risk women: A randomized placebo-controlled double-blind study. Int J Reprod Biomed. 2016 May;14(5):309-16. PMID 27326415
- [Background] Elimian A, Smith K, Williams M, Knudtson E, Goodman JR, Escobedo MB. A randomized controlled trial of intramuscular versus vaginal progesterone for the prevention of recurrent preterm birth. Int J Gynaecol Obstet. 2016 Aug;134(2):169-72. doi: 10.1016/j.ijgo.2016.01.010. Epub 2016 Apr 18. PMID 27168167
- [Background] Conde-Agudelo A, Romero R. Vaginal progesterone to prevent preterm birth in pregnant women with a sonographic short cervix: clinical and public health implications. Am J Obstet Gynecol. 2016 Feb;214(2):235-242. doi: 10.1016/j.ajog.2015.09.102. Epub 2015 Oct 9. PMID 26450404
- [Background] Romero R. Vaginal progesterone to reduce the rate of preterm birth and neonatal morbidity: a solution at last. Womens Health (Lond). 2011 Sep;7(5):501-4. doi: 10.2217/whe.11.60. No abstract available. PMID 21879816
- [Background] Hassan SS, Romero R, Vidyadhari D, Fusey S, Baxter JK, Khandelwal M, Vijayaraghavan J, Trivedi Y, Soma-Pillay P, Sambarey P, Dayal A, Potapov V, O'Brien J, Astakhov V, Yuzko O, Kinzler W, Dattel B, Sehdev H, Mazheika L, Manchulenko D, Gervasi MT, Sullivan L, Conde-Agudelo A, Phillips JA, Creasy GW; PREGNANT Trial. Vaginal progesterone reduces the rate of preterm birth in women with a sonographic short cervix: a multicenter, randomized, double-blind, placebo-controlled trial. Ultrasound Obstet Gynecol. 2011 Jul;38(1):18-31. doi: 10.1002/uog.9017. Epub 2011 Jun 15. PMID 21472815
- [Background] da Fonseca EB, Bittar RE, Carvalho MH, Zugaib M. Prophylactic administration of progesterone by vaginal suppository to reduce the incidence of spontaneous preterm birth in women at increased risk: a randomized placebo-controlled double-blind study. Am J Obstet Gynecol. 2003 Feb;188(2):419-24. doi: 10.1067/mob.2003.41. PMID 12592250
- [Result] Palacio M, Cobo T, Antolin E, Ramirez M, Cabrera F, Mozo de Rosales F, Bartha JL, Juan M, Marti A, Oros D, Rodriguez A, Scazzocchio E, Olivares JM, Varea S, Rios J, Gratacos E; PROMISE Collaborative Group. Vaginal progesterone as maintenance treatment after an episode of preterm labour (PROMISE) study: a multicentre, double-blind, randomised, placebo-controlled trial. BJOG. 2016 Nov;123(12):1990-1999. doi: 10.1111/1471-0528.13956. Epub 2016 Mar 30. PMID 27028759
- [Result] Martinez de Tejada B, Karolinski A, Ocampo MC, Laterra C, Hosli I, Fernandez D, Surbek D, Huespe M, Drack G, Bunader A, Rouillier S, Lopez de Degani G, Seidenstein E, Prentl E, Anton J, Krahenmann F, Nowacki D, Poncelas M, Nassif JC, Papera R, Tuma C, Espoile R, Tiberio O, Breccia G, Messina A, Peker B, Schinner E, Mol BW, Kanterewicz L, Wainer V, Boulvain M, Othenin-Girard V, Bertolino MV, Irion O; 4P trial group. Prevention of preterm delivery with vaginal progesterone in women with preterm labour (4P): randomised double-blind placebo-controlled trial. BJOG. 2015 Jan;122(1):80-91. doi: 10.1111/1471-0528.13061. Epub 2014 Sep 11. PMID 25209926
- [Result] Borna S, Sahabi N. Progesterone for maintenance tocolytic therapy after threatened preterm labour: a randomised controlled trial. Aust N Z J Obstet Gynaecol. 2008 Feb;48(1):58-63. doi: 10.1111/j.1479-828X.2007.00803.x. PMID 18275573
- [Result] Arikan I, Barut A, Harma M, Harma IM. Effect of progesterone as a tocolytic and in maintenance therapy during preterm labor. Gynecol Obstet Invest. 2011;72(4):269-73. doi: 10.1159/000328719. Epub 2011 Nov 12. PMID 22086108